CLINICAL TRIAL: NCT03813615
Title: Preoperative Aerobic Training for Solid Tumors (PRESTO 1): A Phase 0/1a Digitized Clinical Trial
Brief Title: Study of the Effects of Pre-surgical Aerobic Exercise on Patients With Solid Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-534
Record Dates: First submitted 2019-01-21; First posted 2019-01-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Preoperative Aerobic Training; Solid Tumors
Keywords: Aerobic Training; 18-534

STUDY DESIGN:
Intervention Model Description: This protocol is a single-center, open-label, phase 0 / 1 a/b study of preoperative aerobic training in patients with untreated solid tumors. This study design allows for the enrollment of patients with various types of cancer. This study will target patients with prespecified solid malignancies.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot "Proof-of-Concept" (Experimental): Individualized, progressive aerobic training consisting of treadmill walking for a total of 150 mins/wk delivered over 5 sessions/wk following a linear (breast, prostate, and endometrial) or non-linear (lung) dosing schedule for a minimum of 2 weeks.
  Interventions: Behavioral: treadmill walking (Proof-of-Concept)
- Phase 1a: Dose-Finding / Escalation (Experimental): Individualized, progressive aerobic training consisting of treadmill walking ranging from a total of 90 mins/wk to 450 mins/wk delivered over 3 to 7 sessions/wk following a linear or non-linear dosing schedule for a minimum of 2 weeks. If a patient is temporarily unable to complete supervised sessions as a result of unforeseen circumstances, patients may be assigned low intensity unsupervised training sessions per EP/PI discretion.
  Interventions: Behavioral: treadmill walking Dose-Finding / Escalation

INTERVENTIONS:
Behavioral: treadmill walking (Proof-of-Concept) — Individualized, progressive aerobic training consisting of treadmill walking for a total of 150 mins/wk delivered over 5 sessions/wk following a linear dosing schedule for a minimum of 2 weeks. All aerobic training treatment will be implemented and may be monitored using TeleEx. Participants may also perform up to two aerobic training sessions per week in an unsupervised home-based setting. Patients will be provided with Appendix J - Unsupervised Home-Based Exercise Recording Form and Appendix K - Unsupervised Home-Based Exercise Instructions to record their sessions. General physical activity as well as exercise performed outside of the structured treatment sessions will be evaluated via continuous monitoring using MSK approved telemedicine / wireless technology. setting.
  Arms: Pilot "Proof-of-Concept"
Behavioral: treadmill walking Dose-Finding / Escalation — Six doses of aerobic training ( 90mins/wk, 150 mins/wk, 225 mins/wk, 300 mins/wk & 450mins/wk) delivered following either a standard linear (i.e., each dose of exercise is performed at the same intensity & duration) or non-linear (i.e., exercise dose is continually altered & progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule 3 to 6 times weekly (over a 7-day period) for a minimum 2 weeks. Aerobic training treatment will be implemented & may be monitored using TeleEx. Patients may also perform up to three aerobic training sessions per week in an unsupervised home-based setting. Patients will be provided a plan for their unsupervised session(s) verbally or via Portal Secure Messaging (PSM), as appropriate.
  Arms: Phase 1a: Dose-Finding / Escalation

SUMMARY:
The purpose of this study is to find the safest level of aerobic training for people about to undergo surgery for their cancer, and to learn what effects, if any, aerobic exercise has on these patients and the outcomes of their cancers. This part of the study (Phase 0) will evaluate the feasibility and quality of at-home exercise and assessment procedures and find out whether study participants are willing to practice continuous lifestyle monitoring using apps and electronic devices.

Phase 1a will compare the effects and feasibility of six different doses of aerobic exercise and will continue evaluating the quality of at-home study procedures, which includes the use of continuous lifestyle monitoring through apps and electronic devices.

In order to facilitate completion of the phase 1a component, we will backfill the 90, 225, and 300 mins/wk dosing cohorts with at least 4 patients in each dose cohort.

ELIGIBILITY:
Inclusion Criteria:

Phase 0 (Proof-of-Concept)

* Patients with one of the following:

  * Early-stage breast cancer having completed participation in IRB# 15-147
  * Diagnosed with the prespecified solid tumors: endometrial, breast or prostate cancer
  * Underwent a diagnostic lung biopsy within 14 days prior to enrollment
  * Age >18 years
  * BMI ≤ 40
  * Has ≥ 20 mg of fresh normal lung and suspicious lung tissue from the standard of care diagnostic biopsy available for snap freezing and single-cell sequencing (lung patients only)
  * At least a 2-week window from study enrollment to scheduled surgical resection (patients with prespecified solid tumors only)
  * Performing less than 30 minutes of structured moderate-intensity or strenuous-intensity exercise per week, as evaluation by self report If > 30 minutes but less than 90 minutes, patients may be eligible, at the discretion of the PI.
  * Cleared for exercise participation as per screening clearance via PAR-Q+
  * Willingness to comply with all study-related procedures

Phase 1a (Dose-Finding/Escalation)

* Patients with operable untreated prostate cancer scheduled for surgery
* At least a 2-week window from study enrollment to scheduled surgical resection (patients with prespecified solid tumors only)
* Age > 18 years
* BMI </=40
* If BMI >40, patients may be eligible, at the discretion of the PI
* Performing </= 30 minutes of structured moderate-intensity or strenuous-intensity exercise per week, as evaluation by self report If > 30 minutes but less than 90 minutes, patients may be eligible, at the discretion of the PI.
* Cleared for exercise participation as per screening clearance via PAR-Q+
* Willingness to comply with all study-related procedures

Exclusion Criteria:

* Use of any selective estrogen receptor modulator or aromatase inhibitor within 6 months of study entry, including, but not limited to: tamoxifen, raloxifene, arzoxifene, acolbifene, anastrozole, exemestane, and letrozole (for preoperative breast, endometrial, and prostate patients in Phase 0 only)
* Enrollment onto any other interventional investigational study except interventions determined by the PI not to confound the effect of exercise on study outcomes
* Men receiving GNRH agonists and antagonists as well as any antiandrogrens
* Any neoadjuvant anticancer treatment of any kind for the cancer of interest
* Any history of systemic anticancer therapy
* Any other diagnosis of invasive cancer currently requiring active treatment
* Metastatic malignancy of any kind
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the subject a poor candidate for study participation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
identify the recommended dose of aerobic training | 1 year
  The relative dose intensity is defined as the ratio of completed to planned aerobic training dose continually assessed at the end of the intervention period.49 Hence, the maximal feasible dose is defined as the highest dose at which <30% of patients in a dosing cohort fail to achieve the target total cumulative relative dose intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - University of California, Los Angeles (Data Analysis only), Los Angeles, California
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- [Derived] Jones LW, Moskowitz CS, Lee CP, Fickera GA, Chun SS, Michalski MG, Stoeckel K, Underwood WP, Lavery JA, Bhanot U, Linkov I, Dang CT, Ehdaie B, Laudone VP, Eastham JA, Collins A, Sheerin PT, Liu LY, Eng SE, Boutros PC. Neoadjuvant Exercise Therapy in Prostate Cancer: A Phase 1, Decentralized Nonrandomized ControlledTrial. JAMA Oncol. 2024 Sep 1;10(9):1187-1194. doi: 10.1001/jamaoncol.2024.2156. PMID 39023900
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm